CLINICAL TRIAL: NCT07151898
Title: Evaluation of Treatment Response to Trop2 ADC by 68Ga-MY6349 PET/CT in NSCLC
Brief Title: PET/CT for Trop2 ADC Response Evaluation NSCLC
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMYY-2025KY101
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: NSCLC; Trop2; PET/CT
Keywords: NSCLC; Trop2; PET/CT; Trop2-ADC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 68Ga-MY6349 PET/CT: Each participant will receive an intravenous injection of 68Ga-MY6349 and undergo PET/CT imaging at baseline and following two and/or four cycles of Trop2-ADC therapy.
  Interventions: Diagnostic Test: 68Ga-MY6349 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-MY6349 PET/CT — Each participant will receive an intravenous injection of 68Ga-MY6349 and undergo PET/CT imaging at baseline and following two and/or four cycles of Trop2-ADC therapy.

SUMMARY:
To evaluate whether serial 68Ga-MY6349 PET/CT imaging can serve as a noninvasive biomarker to predict the therapeutic efficacy of Trop2-targeted antibody-drug conjugate (Trop2-ADC) therapy in NSCLC patients.

DETAILED DESCRIPTION:
Patients diagnosed with metastatic Non-Small Cell Lung Cancer（NSCLC） will undergo 68Ga-MY6349 PET/CT imaging at baseline and after two and/or four cycles of Trop2-ADC therapy. Tumor uptake will be quantified using both maximum standardized uptake value (SUVmax) and mean SUV (SUVmean). Imaging changes will be correlated with treatment response to assess the utility of 68Ga-MY6349 PET/CT as a predictive biomarker.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or order)
* histologically or cytologically confirmed metastatic NSCLC previously treated with systemic therapy, supported by imaging (e.g. CT, MRI), tumor markers, or pathology reports
* presence of at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
* willingness to undergo serial 68Ga-MY6349 PET/CT scans before and during Trop2-ADC therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Ability to provide written informed consent and, where applicable, assent in accordance with the requirements of the Clinical Research Ethics Committee

Exclusion Criteria:

* Evidence of significantly impaired hepatic or renal function
* Estimated life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with previously treated metastatic NSCLC (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
The predictive value of series 68Ga-MY6349 PET/CT in patients with NSCLC who received Trop2-ADC therapy | 2025.5-2027.5
  For 68Ga-MY6349 PET/CT parameter, the maximum standard uptake value (SUVmax) is measured by defining a region of interest (ROI) around the primary tumor. SUVmax values obtained at baseline and after two and/or four cycles of Trop2-ADC therapy were collected and analyzed in relation to treatment response.

SECONDARY OUTCOMES:
Correlation Between PET Parameters and Survival | 2025.5-2027.5
  Progression-free survival (PFS) amd overall survival (OS) will be monitored and analyzed in relation to imaging parameters obtained from serial 68Ga-MY6349 PET/CT scans.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No